CLINICAL TRIAL: NCT01897454
Title: A Phase II Trial of Preoperative FOLFIRINOX Followed by Gemcitabine Based Chemoradiotherapy in Patients With Borderline Resectable Pancreatic Adenocarcinoma
Brief Title: Gemcitabine Hydrochloride, and Radiation Therapy in Patients With Borderline Resectable Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to slower than anticipated accrual
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-570; NCI-2013-01213 (Registry Identifier: NCI); 12-017; 5P30CA013330-42 (NIH)
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Pancreatic Adenocarcinoma; Stage IIA Pancreatic Cancer; Stage IIB Pancreatic Cancer; Stage III Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fluorouracil; dehydroftorafur; Gemcitabine; Radiotherapy, Intensity-Modulated; Irinotecan; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (FOLFIRINOX, IMRT, and gemcitabine hydrochloride) (Experimental): CHEMOTHERAPY REGIMEN: Patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and irinotecan hydrochloride IV over 90 minutes on day 1, and fluorouracil IV over 46 hours on days 1-3. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients not achieving disease progression proceed to chemoradiotherapy.
  CHEMORADIOTHERAPY REGIMEN: Beginning 4-6 weeks after completion of chemotherapy, patients undergo IMRT on 5 consecutive days per week for a total of 28 fractions and receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, 15, 22, 29, and 36. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fluorouracil; Drug: Gemcitabine Hydrochloride; Radiation: Intensity-Modulated Radiation Therapy; Drug: Irinotecan Hydrochloride; Drug: Leucovorin Calcium; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; Irinomedac; U-101440E
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669

SUMMARY:
This phase II trial studies how well combination chemotherapy, gemcitabine hydrochloride, and radiation therapy before surgery works in treating patients with pancreatic cancer that has not spread to other places in the body and can be removed by surgery. Drugs used in chemotherapy, such as fluorouracil, leucovorin calcium, irinotecan hydrochloride, oxaliplatin, and gemcitabine hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Fluorouracil, irinotecan hydrochloride, and gemcitabine hydrochloride may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving combination chemotherapy and gemcitabine hydrochloride with radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy, measured as the proportion of R0 resections, of fluorouracil-leucovorin calcium-irinotecan hydrochloride-oxaliplatin (FOLFIRINOX) chemotherapy regimen followed by gemcitabine based chemoradiotherapy when used as preoperative therapy in patients with borderline resectable adenocarcinoma of the pancreas.

SECONDARY OBJECTIVES:

I. To measure the overall response rate (ORR). II. To evaluate overall survival (OS). III. To evaluate progression free survival (PFS). IV. To evaluate safety and toxicity associated with chemotherapy and radiotherapy.

V. To assess adverse events related to surgery. VI. To assess the proportion of patients able to undergo resection. VII. To assess proportion of patients requiring vascular reconstruction.

OUTLINE:

CHEMOTHERAPY REGIMEN: Patients receive oxaliplatin intravenously (IV) over 2 hours, leucovorin calcium IV over 2 hours, and irinotecan hydrochloride IV over 90 minutes on day 1, and fluorouracil IV over 46 hours on days 1-3. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients not achieving disease progression proceed to chemoradiotherapy.

CHEMORADIOTHERAPY REGIMEN: Beginning 4-6 weeks after completion of chemotherapy, patients undergo intensity-modulated radiation therapy (IMRT) on 5 consecutive days per week for a total of 28 fractions and receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, 15, 22, 29, and 36. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 30 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas
* Only patients that have not received any prior treatment for pancreas cancer are eligible for this treatment protocol
* Patients are not required to have measurable disease by traditional Response Evaluation Criteria in Solid Tumors (RECIST) criteria, as lesions in the pancreas are notoriously hard to measure radiographically; however, patients must have disease which is evaluable for resection
* Disease should be determined as "borderline resectable" according to the Expert Consensus Statement published by Callery et al:

  * No distant metastasis
  * Venous involvement of the superior mesenteric vein (SMV)/portal vein demonstrating tumor abutment with or without impingement and narrowing of the lumen, encasement of the SMV/portal vein but without encasement of the nearby arteries, or short segment venous occlusion resulting from either tumor thrombus or encasement but with suitable vessel proximal and distal to the area of vessel involvement, allowing for safe resection and reconstruction
  * Gastroduodenal artery encasement up to the hepatic artery with either short segment encasement or direct abutment of the hepatic artery, without extension to the celiac axis
  * Tumor abutment of the superior mesenteric artery (SMA) not to exceed greater than 180 degrees of the circumference of the vessel wall
* Life expectancy of greater than 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 80%)
* Leukocytes >= 3,000/microliter (mcL)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 2 mg/dl
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Ability to understand and the willingness to sign a written informed consent document
* Patients may not be receiving any other concurrent chemotherapy, immunotherapy, or radiotherapy

Exclusion Criteria:

* Patients who have had prior chemotherapy or radiotherapy for the treatment of pancreas cancer
* Patients may not be receiving any other investigational agents
* Evidence of extent of pancreatic cancer beyond that defined as "borderline resectable" above (locally advanced or distant disease); peripancreatic lymph node involvement, either confirmed or suspected, will not be considered distant disease unless the lymph node involvement extends outside of the field of resection
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 5-fluorouracil, oxaliplatin, irinotecan or gemcitabine
* Any concurrent active malignancy other than non-melanoma skin cancers or carcinoma-in-situ of the cervix; patients with previous malignancies but without evidence of disease for > 3 years will be allowed to enter the trial; patients with a history of a T1a or b prostate cancer (detected incidentally at transurethral resection of the prostate [TURP] and comprising less than 5% of resected tissue) may participate if the prostate-specific antigen (PSA) remained within normal limits since TURP removal
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-01-27 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Chuy, Principal Investigator — Montefiore Medical Center-Weiler Hospital
Locations (1):
- Montefiore Medical Center-Weiler Hospital, The Bronx, New York, United States

REFERENCES:
- [Derived] Acuna-Villaorduna A, Shankar V, Wysota M, Jirgal A, Kabarriti R, Bellemare S, Goldman I, Kaubisch A, Aparo S, Goel S, Chuy J. Induction Chemotherapy With FOLFIRINOX Followed by Chemoradiation With Gemcitabine in Patients With Borderline-Resectable Pancreatic Ductal Adenocarcinoma. Cancer Control. 2022 Jan-Dec;29:10732748221134411. doi: 10.1177/10732748221134411. PMID 36221952

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled into the study between 1/27/2012 and 04/24/2019.
Groups:
- Treatment (FOLFIRINOX, IMRT, and Gemcitabine Hydrochloride): CHEMOTHERAPY REGIMEN: Patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and irinotecan hydrochloride IV over 90 minutes on day 1, and fluorouracil IV over 46 hours on days 1-3. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients not achieving disease progression proceed to chemoradiotherapy.
  CHEMORADIOTHERAPY REGIMEN: Beginning 4-6 weeks after completion of chemotherapy, patients undergo IMRT on 5 consecutive days per week for a total of 28 fractions and receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, 15, 22, 29, and 36. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Fluorouracil: Given IV
  Gemcitabine Hydrochloride: Given IV
  Intensity-Modulated Radiation Therapy: Undergo IMRT
  Irinotecan Hydrochloride: Given IV
  Leucovorin Calcium: Given IV
  Oxaliplatin: Given IV
Period: Overall Study
Arm/Group | Treatment (FOLFIRINOX, IMRT, and Gemcitabine Hydrochloride)
Started | 23
Completed | 22
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (FOLFIRINOX, IMRT, and Gemcitabine Hydrochloride)
Number analyzed (Participants) | 22
Age, Continuous [Median (Standard Deviation); unit: years] | 63.5 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 4
  Non-Hispanic Black | 8
  Hispanic/Latino | 10
Region of Enrollment [Number; unit: participants]
  United States | 22
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.3 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving R0 Resection (R0 Resection Rate)
Description: The percentage of participants achieving R0 resection, defined as the absence of gross and microscopic tumor involvement in the resection margins, will be determined for those participants who receive at least one cycle of FOLFIRINOX chemotherapy. A 90% confidence interval will be determined.
Time Frame: Up to 30 months
Population: Analytical results for the 18 participants who completed neoadjuvant (FOLFIRINOX) treatment
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment (FOLFIRINOX, IMRT, and Gemcitabine Hydrochloride)
Number analyzed (Participants) | 18
Percentage of Participants | 55.6 [33.3 to 68.3]

2. Secondary Outcome: Adverse Events Related to Surgery
Description: Adverse events related to surgical resection will be documented and evaluated using the Clavien-Dindo classification scale. The Clavien-Dindo Classification is used to rank the severity of a surgical complication with higher Grades indicative of more intense interventional therapy needed to correct the complication. Scale grades range from Grade I to Grade V. Grade I complications are usually mild and consist of any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological intervention. Grade II complications require pharmacological treatment with drugs other than such allowed for Grade I. Grade III complications require surgical, endoscopic, or radiological intervention, Grade IV are indicative of life-threatening complications requiring ICU management and Grade V signify death of patient.
Time Frame: Up to 30 months
Population: Data related to the number of surgical adverse events was not collected and analyzed for the 15 participants who underwent surgical resection
Arm/Group | Treatment (FOLFIRINOX, IMRT, and Gemcitabine Hydrochloride)
Number analyzed (Participants) | 0

3. Secondary Outcome: Toxicities Associated With Chemotherapy and Radiotherapy
Description: The number of patients who experienced treatment related adverse events will be determined for all patients who received at least one cycle of FOLFIRINOX chemotherapy. These events will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: Up to 30 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (FOLFIRINOX, IMRT, and Gemcitabine Hydrochloride)
Number analyzed (Participants) | 22
Participants | 22

4. Secondary Outcome: Overall Survival (OS)
Description: Median Overall Survival defined as the the duration of time from diagnosis to the time of death from any cause will be determined.
Time Frame: Up to 60 months
Population: Median overall survival was determined for the 15 patients who received preoperative chemoradiotherapy and underwent pancreaticoduodenectomy
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (FOLFIRINOX, IMRT, and Gemcitabine Hydrochloride)
Number analyzed (Participants) | 15
Months | 35.1 [18.4 to 78.5]

5. Secondary Outcome: Overall Response Rate
Description: Overall Response Rate, defined as the percentage of patients that achieved Partial Response (PR) or Complete Response (CR) as per the Response evaluation in solid tumors criteria, was assessed using RECIST Version 1.1 criteria. Complete Response (CR) is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR) is defined as having at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Higher percentages of PR and CR are associated with more favorable outcomes
Time Frame: Up to 30 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (FOLFIRINOX, IMRT, and Gemcitabine Hydrochloride)
Number analyzed (Participants) | 22
Participants | 4

6. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free Survival defined as the duration of time from start of treatment to time of disease progression will be analyzed. Median progression free survival will be presented.
Time Frame: From start of treatment to time of progression, assessed up to 60 months
Population: as for outcome 4
Measure: Median (Standard Error); unit: Months
Arm/Group | Treatment (FOLFIRINOX, IMRT, and Gemcitabine Hydrochloride)
Number analyzed (Participants) | 15
Months | 34 (9.81)

7. Secondary Outcome: Percentage of Patients Able to Undergo Resection
Description: The percentage of participants with resectable or borderline resectable disease to undergo resection will be determined. The ability for patients to complete preoperative therapy and undergo resection is correlated with more favorable overall survival outcomes.
Time Frame: Up to 30 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (FOLFIRINOX, IMRT, and Gemcitabine Hydrochloride)
Number analyzed (Participants) | 22
Participants | 15

8. Secondary Outcome: Vascular Reconstruction
Description: The percentage of patients who underwent pancreaticoduodenectomy requiring vascular reconstruction will be evaluated.
Time Frame: Up to 30 months
Population: 15 participants underwent pancreaticoduodenectomy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (FOLFIRINOX, IMRT, and Gemcitabine Hydrochloride)
Number analyzed (Participants) | 15
Participants | 5

ADVERSE EVENTS:
Time Frame: Up to 2-6 weeks following each cycle of chemoradiotherapy, up to 60 months
Arm/Group | Treatment (FOLFIRINOX, IMRT, and Gemcitabine Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 1/22
Serious Adverse Events (participants affected / at risk) | 4/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (FOLFIRINOX, IMRT, and Gemcitabine Hydrochloride) (N=22)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) — Verbatim term
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (FOLFIRINOX, IMRT, and Gemcitabine Hydrochloride) (N=22)
Neutropenia (Blood and lymphatic system disorders) | 19 — Verbatim term
Thrombocytopenia (Blood and lymphatic system disorders) | 20 — Verbatim term
Anemia (Blood and lymphatic system disorders) | 10
Fatigue (General disorders) | 19
Nausea (Gastrointestinal disorders) | 11
Diarrhea (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 6
Mucositis (Gastrointestinal disorders) | 5 — Verbatim term
Hand-foot Syndrome (Infections and infestations) | 1 — Verbatim term

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT01897454/Prot_SAP_000.pdf